CLINICAL TRIAL: NCT04328363
Title: Social Prescription of Health Assets and Lifestyles Modification by Primary Care Nurses to Reduce Glycemia in People With Prediabetes: PREDIBAL Study -a Cluster-randomized Hybrid Effectiveness-implementation Type II Trial Protocol
Brief Title: Social Prescription and Lifestyles Modification to Reduce Glycemia in People With Prediabetes (PREDIBAL)
Acronym: PREDIBAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of the Balearic Islands (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PREDIBAL
Record Dates: First submitted 2020-03-27; First posted 2020-03-31 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: PreDiabetes
MeSH Terms: conditions — Prediabetic State | interventions — Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention will be carried out by primary care nurses over eight visits: baseline visit and follow-up visits which take place 15 days, 1, 2, 4, 6, 9, and 12 months after baseline with a final visit evaluation at 18 months. The intervention will be based on the social prescription of health assets related to the practice of physical activity and a healthy eating pattern to modify lifestyles in people with prediabetes. The content of the intervention proposed is based on the NHS and it will be carried out at three levels (individual, group and community) to facilitate the patient empowerment and promotion of healthy lifestyles with a positive orientation using the community resources.
  Interventions: Behavioral: Intervention
- Control (No Intervention): The Control group will receive routine standard care.

INTERVENTIONS:
Behavioral: Intervention — Social prescription of health assets related to the practice of physical activity and a healthy eating pattern to modify lifestyles.
  Arms: Intervention

SUMMARY:
This study aims to evaluate the effectiveness and cost-utility of an intervention based on the social prescription of health assets to modify lifestyles and reduce blood glucose values in prediabetic patients in primary care nursing consultations.

Multicentre, controlled and randomized (two different branches) clinical trial with 18 months of follow-up will be performed. The intervention group will receive a social prescription of health assets related to the practice of physical activity and healthy eating patterns in primary care nursing consultation.

DETAILED DESCRIPTION:
No pragmatic clinical trial evaluating the effectiveness of prevention interventions has been performed to date. Social prescription is a useful health promotion strategy that facilitates the continuity of individual care. This randomized controlled trial aims to evaluate the effectiveness and cost-utility of an intervention based on the social prescription of health assets to modify lifestyles and reduce blood glucose values in prediabetic patients in primary care nursing consultations. Additional aims are to describe and assess barriers, motivations, and attitudes of patients with low adherence to the intervention and their association with social class and gender.

Methods: Multicentre, controlled and randomized (two different branches) clinical trial with 18 months of follow-up will be performed. The randomization unit will be the primary healthcare center. The study will be conducted by nurses in 12 primary health care centers (PHC) of Mallorca in Spain that will be included and randomly allocated to intervention or control groups. Furthermore, the intervention will be delivered at the PHC level, which is considered the unit of analysis. At least 232 patients (116 per branch) will be recruited. Participants will be aged 25 to 75 years with altered fasting glucose levels (100-125 mg/dl) or with glycosylated hemoglobin (HbA1c) between 5.7 and 6.4%. The intervention will be carried out at three levels: community, group and individually. The intervention group will receive a social prescription of health assets related to the practice of physical activity and healthy eating patterns in primary care nursing consultation for 8 sessions during 12 months of follow-up. The Control group will follow the usual care recommendations. Data will be collected at baseline, 6, 12 and 18 months. Glycaemia, HbA1c, BMI and waist circumference will be measured, as well as the Mediterranean diet adherence (PREDIMED), the physical activity (IPAQ), the cardiovascular risk (REGICOR equation), the quality of life (EuroQoL-5D), the social class, gender, and financial costs.

.

ELIGIBILITY:
Inclusion Criteria:

* Fasting basal blood glucose levels between 100 and < 126 mg/dl or HbA1c between 5.7 - 6.4%

Exclusion Criteria:

* Patients with T2D or in treatment with oral antidiabetic drugs
* Institutionalized patients
* Terminal illness, dementia or cognitive impairment;
* Pregnancy
* Surgery or hospital admission in the previous 3 months
* Hematological diseases that could interfere in HbA1c determination
* Presence of any condition that limits the participation in the study
* Participation in a clinical trial or receive a social prescription of diet or physical activity.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Glucosa level | 18 month
  The primary outcome will be the percentage of participants reducing at least 4 mg/dl of FPG

SECONDARY OUTCOMES:
Reversion to normal glucose | 18 month
  Percentage of patients who reverse to normal glucose levels

CONTACTS AND LOCATIONS:
Overall Officials: Miquel Bennasar, PhD, Principal Investigator — University of balearic islands

IPD SHARING:
Plan to Share IPD: No